CLINICAL TRIAL: NCT03813160
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 3 Trial to Evaluate Efficacy and Safety of Lenabasum in Dermatomyositis
Brief Title: Trial to Evaluate Efficacy and Safety of Lenabasum in Dermatomyositis
Acronym: DETERMINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corbus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JBT101-DM-002
Record Dates: First submitted 2019-01-21; First posted 2019-01-23 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Dermatomyositis
Keywords: dermatomyositis; cannabinoid receptor type 2 agonist; JBT-101; lenabasum
MeSH Terms: conditions — Dermatomyositis | interventions — lenabasum; anabasum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lenabasum 20 mg (Experimental): Subjects will receive lenabasum 20 mg twice daily
  Interventions: Drug: Lenabasum 20 mg
- Lenabasum 5 mg (Experimental): Subjects will receive lenabasum 5 mg twice daily
  Interventions: Drug: Lenabasum 5 mg
- Placebo (Placebo Comparator): Subjects will receive placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lenabasum 20 mg — oral capsule
  Other Names: JBT-101; anabasum
  Arms: Lenabasum 20 mg
Drug: Lenabasum 5 mg — oral capsule
  Other Names: JBT-101; anabasum
  Arms: Lenabasum 5 mg
Drug: Placebo — oral capsule
  Arms: Placebo

SUMMARY:
This is a Phase 3 multicenter, double-blind, randomized, placebo-controlled study assessing the efficacy and safety of lenabasum for the treatment of dermatomyositis. Approximately 150 subjects will be enrolled in this study at about 60 sites in North America, Europe, and Asia. The planned duration of double-blind treatment with study drug is up to 52 weeks.

DETAILED DESCRIPTION:
Subjects will be randomized to receive lenabasum 20 mg twice per day, lenabasum 5 mg twice per day, or placebo twice per day in a 2:1:2 ratio. The primary efficacy outcome at Week 28 will compare lenabasum 20 mg BID to placebo the Total Improvement Score (TIS), which is a weighted composite measure of improvement from baseline in six endpoints: Physician Global Assessment of Disease Activity, Physician Assessment of Extramuscular Disease Activity, Patient Global Assessment of Disease Activity, Health Assessment Questionnaire (patient-reported disability), Manual Muscle Testing (MMT), and muscle enzymes.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill at least one of the following criteria for dermatomyositis:

  1. Bohan and Peter criteria (Bohan and Peter, 1975a; Bohan and Peter 1975b)
  2. ACR/EULAR criteria (Lundberg et al, 2017)
* Disease activity/severity fulfills at least one of the following three criteria:

  1. MDGA ≥ 3 cm (0 - 10 cm Visual Analog Scale [VAS]) and MMT-8 score ≤ 142 (out of 150 total possible)
  2. Sum of MDGA, PtGA and EMGA VAS scores is ≥ 10 cm (0-10 cm VAS for each)
  3. MDGA ≥ 3 cm (0-10 cm VAS) and CDASI activity score of > 14
* Stable doses of immunosuppressive medications for DM as defined by:

  1. Unchanged dose of oral corticosteroids ≤ 20 mg per day prednisone or equivalent for ≥ 4 weeks before Visit 1
  2. Unchanged dose of immunosuppressive medications other than oral corticosteroids for ≥ 8 weeks before Screening

Exclusion Criteria:

* Unstable DM or DM with end-stage organ involvement at Screening or Visit 1
* Significant diseases or conditions other than DM that may influence response to the study drug or safety
* Any of the following values for laboratory tests at Screening:

  1. A positive pregnancy test (or at Visit 1)
  2. Hemoglobin < 9 g/dL in males and < 8 g/dL in females
  3. Neutrophils < 1.0 × 10^9/L
  4. Platelets < 75 × 10^9/L
  5. Creatinine clearance < 50 mL/min on screening blood test, per the Modification of Diet in Renal Disease Study or in 24 hour urine creatine clearance measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Efficacy of lenabasum 20 mg BID compared to placebo BID as measured by Total Improvement Score (TIS) | Week 28
  TIS from IMAC Core Set Measures (CSM) will be calculated following Aggarwal et al (2017) recommendations. Scores are based on a 0 - 100 scale; higher scores indicate better improvement in myositis.

SECONDARY OUTCOMES:
Subjects who achieve Definition of Improvement (DOI) | Week 28
  Defined as ≥ 3 of 6 core set measures improved by ≥ 20% (relative to Baseline) with no more than 2 core set measures worsening by ≥ 25% (MMT-8 may not decrease by ≥ 25% from baseline)
Subjects who improve by at least one category on the Investigator Global Assessment (IGA) scale of skin activity | Week 28
  The IGA is used by the investigator to score overall skin disease on a 0 to 4 scale; higher scores indicate greater skin disease.
Change in Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) activity score | Week 28
  CDASI is a validated outcome measure that systematically quantifies cutaneous DM disease activity and damage (Klein et al, 2007; Yassaee et al, 2010) Disease Activity Score is rated using three activity measures. The activity score ranges from 0 to 100. Higher scores indicate greater disease severity.
Subjects who achieve TIS >= 40 (at least moderate improvement) | Week 28
  TIS from IMAC Core Set Measures (CSM) will be calculated following Aggarwal et al (2017) recommendations. Scores are based on a 0 - 100 scale; higher scores indicate better improvement in myositis.
TIS in subjects receiving immunosuppressive therapies (including corticosteroids) for > 1 year at Baseline | Week 52
  TIS from IMAC Core Set Measures (CSM) will be calculated following Aggarwal et al (2017) recommendations. Scores are based on a 0 - 100 scale; higher scores indicate better improvement in myositis.
Change in Forced vital capacity (FVC) absolute, in all subjects and those with interstitial lung disease (ILD) at Baseline. | Week 28
  ILD is defined as a history of fibrosis on chest x-ray, a history of ILD on CT of lungs, and/or FVC% predicted <80% at Screening or Visit 1
Change in Forced vital capacity (FVC) percent predicted, in all subjects and those with interstitial lung disease (ILD) at Baseline. | Week 28
  ILD is defined as a history of fibrosis on chest x-ray, a history of ILD on CT of lungs, and/or FVC% predicted <80% at Screening or Visit 1
TIS at Visit 10 | Week 52
  TIS from IMAC Core Set Measures (CSM) will be calculated following Aggarwal et al (2017) recommendations. Scores are based on a 0 - 100 scale; higher scores indicate better improvement in myositis.
TIS, lenabasum 5 mg BID versus placebo | Week 28
  TIS from IMAC Core Set Measures (CSM) will be calculated following Aggarwal et al (2017) recommendations. Scores are based on a 0 - 100 scale; higher scores indicate better improvement in myositis.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria P Werth, MD, Principal Investigator — University of Pennsylvania; Chester V Oddis, MD, Principal Investigator — University of Pittsburgh Department of Medicine/Division of Rheumatology
Locations (54):
- United States (23):
  - HonorHealth Neurology, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Attune Health Center, Beverly Hills, California
  - UCLA Division of Rheumatology, Los Angeles, California
  - Denver Arthritis Clinic, Denver, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - DelRicht Research, New Orleans, Louisiana
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Division of Rheumatic and Autoimmune Diseases, Minneapolis, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Hospital for Special Surgery, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Division of Rheumatology, Pittsburgh, Pennsylvania
  - MUSC: Department of Neurology, Charleston, South Carolina
  - Austin Neuromuscular Center, Austin, Texas
  - Rheumatic Disease Center, Glendale, Wisconsin
- Bulgaria (3):
  - University Hospital "Kaspela" Rheumatology Clinic, Plovdiv
  - UMHAT "St. Ivan Rilski", Sofia
  - UMHAT, Stara Zagora
- University of British Columbia, Dept. of Dermatology and Skin Science, Vancouver, British Columbia, Canada
- Revmatologicky ustav, Prague, Czechia
- Germany (3):
  - Charite-Universitatsmedizin, Berlin
  - University Hospital Erlangen Nuremberg, Erlangen
  - University Medical Center Goettingen, Göttingen
- University of Debrecen, Debrecen, Hungary
- Italy (2):
  - University Hospital Policlinico-Vittorio Emanuele, Catania
  - Fondazione Policlinico Universitario A.Gemelli-IRCCS, Roma
- Japan (9):
  - Gunma University Hospital, Gunma
  - Hokkaido University Hospital, Hokkaido
  - Yokohama City University Hospital, Kanagawa
  - Kyoto University Hospital, Kyoto
  - Tohoku University Hospital, Miyagi
  - Osaka University Hospital, Osaka
  - Keio University Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - Wakayama Medical Hospital, Wakayama
- Poland (3):
  - KLIMED, Bialystok
  - Kliniczny Szpital Wojewodzki Nr 1. im Fryderyka Chopina Klinika Dermatologii, Rzeszów
  - KLIMED, Łomża
- South Korea (4):
  - Inha University Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
- Spain (2):
  - Vall d'Hebron General Hospital, Barcelona
  - Hospital 12 Octubre, Madrid
- Karolinska University Hospital, Rheumatology Clinic, Stockholm, Sweden
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kodali N, Diaz D, Dhiman R, Vazquez T, Feng R, Patel J, Dan J, Sprow G, Kleitsch J, Sharma M, Bashir M, Werth VP. Diverse Lenabasum pathway activation in dermatomyositis patients' blood. Sci Rep. 2025 May 18;15(1):17232. doi: 10.1038/s41598-025-92001-z. PMID 40383862

DOCUMENTS (2):
  • Study Protocol (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/60/NCT03813160/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT03813160/SAP_001.pdf